CLINICAL TRIAL: NCT02220855
Title: A Phase II Study of BKM120 (Buparlisib) in Relapsed or Refractory Thymomas
Brief Title: A Study of BKM120 (Buparlisib) in Relapsed or Refractory Thymomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Joseph Loehrer Sr. (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Patrick Joseph Loehrer Sr., Associate Dean for Cancer Research, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0478
Record Dates: First submitted 2014-08-07; First posted 2014-08-20 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Thymoma
MeSH Terms: conditions — Thymoma | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BKM120 (Experimental): BKM120, 100mg capsule for oral use, taken once daily for two or more months for a maximum of one year. Each cycle is 28 days.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120

SUMMARY:
Thymic tumors are rare tumors, but represent the most common tumors of the anterior mediastinum. Thymoma has an indolent course in advanced disease and has the propensity to spread to the pleura. In first line therapy, combination chemotherapy produces responses in approximately 80% of patients. A number of single agents have activity in recurrent disease, but none are curable. Patients with recurrent thymoma have limited treatment options, and thus novel target modalities are needed.

At the Indiana University Simon Cancer Center (IUSCC), more patients with advance thymoma are seen than any other institution in the country. Our main hypothesis is the PI3K pathway is an important driver for growth and metastasis of thymoma and that inhibition of the PI3K pathway is expected to produce clinically meaningful response in patients with recurrent thymoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of thymoma.
2. At least one prior line of platin-based chemotherapy (unless refused or not tolerated).
3. Documented progressive (clinical and/or objective) disease after the most recent systemic therapy regimen.
4. Patients must not have received chemotherapy, radiation therapy, or undergone major surgery within 4 weeks prior to enrollment.
5. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 4 for the evaluation of measurable disease.
6. Age ≥ 18 years
7. ECOG performance status £ 2
8. Patient must be able to swallow and retain oral medications
9. Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
10. Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
11. Magnesium ≥ the lower limit of normal
12. Potassium within normal limits for the institution
13. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or ≤ 3.0 x upper limit of normal (ULN) if liver metastases are present)
14. Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
15. Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
16. Serum amylase ≤ ULN
17. Serum lipase ≤ ULN
18. Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
19. HbA1c ≤ 8 %
20. Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
21. Signed informed consent
22. INR ≤ 2

Exclusion Criteria:

1. Patients who have received prior treatment with a P13K inhibitor.
2. Patients with thymic carcinoma (formerly WHO Type C).
3. Patients with a known hypersensitivity to BKM120 or to its excipients
4. Patients with untreated brain metastases are excluded. However, patients with metastatic CNS tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (incl. radiation and/or surgery), is clinically stable at the time of study entry and is receiving low dosage corticosteroid therapy
5. Patients with acute or chronic liver, renal disease or pancreatitis
6. Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire: • Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.

   * ≥ CTCAE grade 3 anxiety
   * Meets the cut-off score of ≥ 12 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
7. Patients with diarrhea ≥ CTCAE grade 2
8. Patient has known active cardiac disease including any of the following:

   • Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)
   * QTc > 480 msec on screening ECG (using the QTcF formula)
   * Angina pectoris that requires the use of anti-anginal medication
   * Ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Valvular disease with document compromise in cardiac function
   * Symptomatic pericarditis
9. Patient has a history of cardiac dysfunction including any of the following:

   • Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
   * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Documented cardiomyopathy
10. Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
11. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection; uncontrolled hypertension) that could cause unacceptable safety risks or compromise compliance with the protocol • Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates.
12. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
13. Patients who have been treated with any hematopoietic colony stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
14. Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to table 4 8 or a list of prohibited QT prolonging drugs with risk of Torsades de Pointes.
15. Patients receiving chronic treatment with steroids or another immunosuppressive agent. • Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients with previously treated brain metastases, who are on stable low dose corticosteroid treatment (e,g dexamethasone 2 mg/day, predisolone 10 mg/day) for at least 14 days before start of study treatment are eligible.
16. Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
17. Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Table 4-7 for a list of prohibited inhibitors and inducers of CYP3A (Please note that co-treatment with weak inhibitors of CYP3A is allowed).
18. Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a grade 1 before starting the trial
19. Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half-lives prior to starting study drug or who have not recovered from side effects of such therapy
20. Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
21. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
22. Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
23. Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 72 hours prior to initiating treatment.

    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL [for US only: and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
    * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment for 4 weeks (5 T1/2) (after stopping treatment... The highly effective contraception is defined as either:

1. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

2. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.

3. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that patient.

4. Use of a combination of any two of the following (a+b):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

   * Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.
   * Fertile males, defined as all males physiologically capable of conceiving offspring must use condoms during treatment, for 4 weeks (5 T1/2) after stopping treatment and for an additional 12 weeks (1616 weeks in total after study drug discontinuation) and should not father a child in this period.
   * Female partner of male study subject should use highly effective contraception during dosing of any study agent and for 16 weeks after final dose of study therapy.

     24. Known diagnosis of human immunodeficiency virus (HIV) infection 25. History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix 26. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Loehrer, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Abu Zaid MI, Radovich M, Althouse S, Liu H, Spittler AJ, Solzak J, Badve S, Loehrer PJ Sr. A phase II study of buparlisib in relapsed or refractory thymomas. Front Oncol. 2022 Oct 18;12:891383. doi: 10.3389/fonc.2022.891383. eCollection 2022. PMID 36330484
- [Derived] Radovich M, Solzak JP, Hancock BA, Conces ML, Atale R, Porter RF, Zhu J, Glasscock J, Kesler KA, Badve SS, Schneider BP, Loehrer PJ. A large microRNA cluster on chromosome 19 is a transcriptional hallmark of WHO type A and AB thymomas. Br J Cancer. 2016 Feb 16;114(4):477-84. doi: 10.1038/bjc.2015.425. Epub 2016 Jan 14. PMID 26766736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on enrolling at least 16 patients. The protocol enrolled 14 patients due to lack of funding.
Period: Overall Study
Arm/Group | BKM120
Started | 14
Completed | 0
Not Completed | 14
Not completed — Adverse Event | 8
Not completed — Disease Progression | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | BKM120
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Objective Response
Description: Percent of patients with Objective response and the Binomial Exact 95% confidence interval. Objective response is defined as having a best response of Complete Response (defined as disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10mm) or Partial Response (defined as at least a 30% decrease in the sum of diameters of target lesions from the baseline sum diameters) by RECIST v1.1 criteria.
Time Frame: up to three years
Population: All patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKM120
Number analyzed (Participants) | 14
percentage of participants | 7.1 [0.2 to 33.9]

2. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Above
Description: Number of unique patients who had a treatment related (possible, probable or definite) adverse events with grade >= 3.
Time Frame: up to three years
Population: All patients enrolled and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | BKM120
Number analyzed (Participants) | 14
Participants | 7

3. Secondary Outcome: Progression-free Survival Rate
Description: Duration of time from the start of treatment to time of documented progression or death. Patients who do not progress or die will be censored on their last evaluation date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: up to three years
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM120
Number analyzed (Participants) | 14
months | 11.1 [2.9 to 18.8]

4. Secondary Outcome: Percent of Patients Achieving Disease Control
Description: Percent of patients achieving disease control and the Binomial Exact 95% confidence interval. Disease control is defined as having a best response of Complete Response (defined as disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10mm) or Partial Response (defined as at least a 30% decrease in the sum of diameters of target lesions from the baseline sum diameters) or Stable Disease for at least 4 months (defined by neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progression) by RECIST v1.1 criteria.
Time Frame: up to three years
Population: All patients enrolled and received treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKM120
Number analyzed (Participants) | 14
percentage of participants | 50.0 [23.0 to 77.0]

5. Secondary Outcome: Overall Survival Rate
Description: Duration of time from the start of treatment to time of death due to any causes. Patients who do not die will be censored on their last known alive date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: up to three years
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BKM120
Number analyzed (Participants) | 14
months | 22.5 [10.7 to 31.3]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | BKM120
All-Cause Mortality (participants affected / at risk) | 5/14
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=14)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BKM120 (N=14)
Middle ear inflammation (Ear and labyrinth disorders) | 1
Endocrine disorders - Other (Endocrine disorders) | 2
Cataract (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 11
Fever (General disorders) | 3
Non-cardiac chest pain (General disorders) | 5
Pain (General disorders) | 2
Bronchial infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 3
Lung infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 8
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Psychiatric disorders - Other (Psychiatric disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash acneiform (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT02220855/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT02220855/SAP_001.pdf